CLINICAL TRIAL: NCT01596296
Title: Foley Catheter Versus Dinoprostone Vaginal Insert for Induction of Labor in Parous Women at Term: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FCB_PG_parous women
Record Dates: First submitted 2012-05-09; First posted 2012-05-10 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2016-10

CONDITIONS: Failed Induction of Labor
Keywords: labor induction; transcervical foley catheter; dinoprostone; parous women
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcervical foley catheter (Active Comparator)
  Interventions: Device: Transcervical foley catheter
- Dinoprostone (Active Comparator)
  Interventions: Drug: Dinoprostone 10mg

INTERVENTIONS:
Device: Transcervical foley catheter — 16 French foley catheter insertion
  Arms: Transcervical foley catheter
Drug: Dinoprostone 10mg — Dinoprostone vaginal insertion
  Arms: Dinoprostone

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of transcervical foley catheter as compared to dinoprostone vaginal insertion for preinduction cervical ripening and labor induction in term parous women with unfavorable cervix.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* parous women
* gestational age >=37.0 weeks
* Bishop score <=5
* intact amniotic membrane
* absence of labor
* live fetus with vertex presentation
* no previous uterine surgical procedure

Exclusion Criteria:

* major congenital anomaly

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2012-05; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Successful labor induction | Twelve hours of initiating oxytocin on the first day of induction
  Successful labor induction is defined as an ability to achieve the active phase of labor corresponding to a cervical dilatation of >=4cm.

SECONDARY OUTCOMES:
Cervical change in the bishop scores and cervical lengths induced by transcervical foley catheter and dinoprostone vaginal insertion | When transcervical foley catheter or dinoprostone was removed before adminitoring oxytocin
  1. Cervical change based on the bishop score and cervical length induced by cervical ripening methods(foley catheter balloon vs dinoprostone)
  2. Incidence of cesarean delivery
  3. Vaginal delivery with 24 hours of starting of induction
  4. The interval from start of oxytocin to delivery
  5. Incidence of admission to neonatal intensive care unit and uterine tachysystole

CONTACTS AND LOCATIONS:
Overall Officials: Kyo Hoon Park, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Department of Obstetrics and Gynecology Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264